CLINICAL TRIAL: NCT04821375
Title: Pilot Study of Effects of Bazedoxifene Plus Conjugated Estrogen on Imaging and Blood Biomarkers In Women With Menopausal Symptoms at Increased Risk for Breast Cancer
Brief Title: Pilot Study of Bazedoxifene Plus Conjugated Estrogen on Imaging and Blood Biomarkers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study00146761
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Increased Risk for Development of Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Intervention Model Description: Randomized at enrollment to either immediate study agent or study agent after a 6-months wait.
Masking Description: Only a designated biostatistician and investigational pharmacy personnel will be aware randomization until after a subject is enrolled, and then all involved in the study will be aware of assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bazedoxifene plus conjugated estrogens immediately (Experimental): Immediate receipt of 6 months of bazedoxifene (20 mg) and conjugated estrogens (0.45 mg) taken together daily.
  Interventions: Drug: bazedoxifene plus conjugated estrogens
- Bazedoxifene plus conjugated estrogens wait list (Other): After a 6-month waiting period, receipt of 6 months of bazedoxifene (20 mg) and conjugated estrogens (0.45 mg) taken together daily.
  Interventions: Drug: bazedoxifene plus conjugated estrogens

INTERVENTIONS:
Drug: bazedoxifene plus conjugated estrogens — 6 months of bazedoxifene (20 mg) and conjugated estrogens (0.45 mg) taken together daily.
  Other Names: BZA+CE

SUMMARY:
Pilot study to test feasibility of 6 months of bazedoxifene (BZA) plus conjugated estrogens (CE) to modulate breast MRI parameters.

DETAILED DESCRIPTION:
Duavee® which is the combination of the selective estrogen receptor modulator (SERM) bazedoxifene plus conjugated estrogens is an FDA approved drug for treatment of hot-flashes and prevention of osteoporosis in postmenopausal women. In a single arm pilot study 6 months of Duavee® was associated with improvement in several risk biomarkers including benign breast tissue proliferation, mammographic fibroglandular volume, and progesterone in women in late menopause transition and at high risk for development of breast cancer. Prior to opening a planned randomized Phase IIB trial of 6 months of Duavee® vs placebo in high risk women with hot-flashes followed by open label Duavee®, a pilot trial was initiated of 6 months of Duavee® vs wait-list control in symptomatic women (Study00145121; NCT04379024). This trial was also intended to provide additional imaging biomarker information from MRI which was not performed in the previous prior study. A finding on MRI of greater background parenchymal enhancement (BPE) in high risk women is positively associated with higher probability of developing breast cancer and is independent of fibroglandular volume. BPE is reduced by selective estrogen receptor modulators including tamoxifen. Change in MRI BPE over time was also investigated for women randomly assigned to either receive Duavee® or not (wait-list control), as well as exploration of fully automated breast MRI volumetric density measures.

Unfortunately, midway through the trial, Duavee® became no longer available due to an issue with packaging and dissolution of the active agents. As an alternative, this current protocol will utilize separate agents of bazedoxifene (as Vivant® available from Japan) plus conjugated estrogens (available in the US as Premarin®). The specific objectives are identical to those in Study00145121, with the exception that Duavee® has been replaced by BZA+CE. The intent is to combine the results of both trials for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women who report vasomotor symptoms (hot flashes or night sweats or both).
* No menstrual periods for at least 60 days.
* Age 45-65. Women age 45-49 with prior hysterectomy or endometrial ablation with rare or no periods due to ablation must have a Follicle Stimulating Hormone (FSH) of 25 mIU/ml or higher to be eligible.
* BMI <36 kg/m2
* Risk Factors/Level. Moderate risk of developing breast cancer based on either by having any one or more of the following:

  * First or 2nd degree relative with breast cancer
  * Known carrier of moderate to high penetrance germline mutation
  * Prior breast biopsy showing proliferative breast disease or multiple prior biopsies
  * High mammographic density (Volpara® categories c or d or BIRADS density assessment as heterogeneously or extremely dense (c or d).
  * IBIS Breast Cancer Risk Evaluation Version 8 (http://www.emstrials.org/riskevaluator/). 10-year relative risk of >2X that for the population for age group.
* Prior mammogram must have at least a Volpara® fibroglandular volume of 80 cm3 or BIRADs b, c, or d category density and/or investigator estimated visual dense area of at least 25%. The entire breast must be incorporated in a single view for both the right and left breast. (i.e., women whose breasts are so large that the images must be captured as a mosaic are not eligible). If no prior mammogram, but breast density is readily appreciated and documented on physical exam, a study-provided 3D mammogram with Volpara® software must be performed to document above eligibility criterion. It will then constitute the baseline mammogram.
* Willing to comply with study procedures:

  * Have blood drawn for screening tests - comprehensive metabolic panel (plus FSH if age 45-49 and no uterus or endometrial ablation)
  * Have blood drawn to archive serum for assay of estradiol, testosterone, progesterone, sex hormone binding globulin (SHBG), FSH at baseline and 6-month visits (and 12 months for women originally randomized to wait list control and subsequently taking BZA+CE for the next 6 months).
  * Undergo a history, physical, and breast exam at baseline and 6-month visits (and 12 months for women originally randomized to wait list control and subsequently taking BZA+CE for the next 6 months). History, physical exam and breast exam performed by a study-associated clinician within 3 months prior to enrollment may be substituted for baseline evaluations.
  * Have a mammogram at University of Kansas Medical Center (KUMC) with Volpara® volumetric density at baseline and 6-month visits (and 12 months for women originally randomized to wait list control and subsequently taking BZA+CE for the next 6 months).
  * Have a study provided abbreviated MRI at KUMC at baseline and 6-month visits.
  * Be contacted by the trial coordinator by phone, email, or text at months 1 and 3 (and months 7 and 9 for women originally randomized to wait list control and subsequently taking BZA+CE for the next 6 months).
  * Complete Mayo Clinic hot flash assessment at baseline and 6-month visits (and month 12 for women originally randomized to wait list control and subsequently taking BZA+CE for the next 6 months).
  * Women 45-55 with a functional uterus (e.g., no prior endometrial ablation), menstrual period in the past 12 months, and heterosexually active, must be agreeable to use some non-hormonal form of contraception while taking BZA+CE unless husband or partner has had a vasectomy.
* Able to understand and sign an informed consent form for screening and for intervention.
* Participants on the optional random periareolar fine needle aspiration (RPFNA) procedures must meet eligibility criteria for participation on HSC4601, Breast Random Fine Needle Aspiration and/or Nipple Aspirate Fluid Collection of Breast Tissue to Aid in Short-term Risk Assessment. Participants must sign a separate optional consent for this study as well as for HSC4601. However, any eligibility criteria dealing with hormone replacement therapy and SERMs are excluded to allow the 6-month aspiration.
* Comprehensive Metabolic Panel shows clinically acceptable renal and hepatic function lab values.
* For women with intact uterus and ovary(ies) and less than age 55, a negative pregnancy test is required.

Exclusion Criteria:

* Risk: A prior biopsy showing pleomorphic lobular or ductal carcinoma in situ or invasive breast cancer.
* Medical Conditions:

  * Have a predisposition to or prior history of thromboembolism, deep venous thrombosis, pulmonary embolism, or stroke
  * History of renal or liver disease
  * Prior invasive ovarian or endometrial cancer
  * Any other condition or intercurrent illness that in the opinion of the investigator makes the woman a poor candidate for BZA+CE.
* Medications

  * Taking systemic hormones within two months (eight weeks) prior to baseline MRI and mammogram.
  * Taking systemic hormones within two months (eight weeks) prior to baseline MRI and mammogram.
  * Taking tamoxifen, raloxifene, Duavee®, or any selective estrogen receptor modulator, or an aromatase inhibitor within 12 months prior to baseline MRI and mammogram.

Exclusion Criteria after baseline studies:

* Mammogram with Volpara® software and/or abbreviated MRI interpreted as concerning for cancer - unless recommended breast biopsy has been performed and confirmed as benign.
* Dispensing of BZA+CE for those randomized to receive it immediately does not occur within 3 months of baseline MRI.
* Unwilling to comply with future study procedures.
* Started hormone replacement, selective estrogen receptor modulator, or aromatase inhibitor after baseline studies performed but prior to randomization.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of potential participants who consent to enrollment | Enrollment
  Trial design is acceptable to potential subjects, as evidenced by participation

SECONDARY OUTCOMES:
Change in breast background parenchymal enhancement (BPE) | 6 months
  BPE assessed by abbreviated MRI at baseline and after 6 months
Change in fibroglandular volume (FGV) | 6 months
  FGV assessed by Volpara software on 3D mammograms acquired at baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabian CJ, Nye L, Powers KR, Nydegger JL, Kreutzjans AL, Phillips TA, Metheny T, Winblad O, Zalles CM, Hagan CR, Goodman ML, Gajewski BJ, Koestler DC, Chalise P, Kimler BF. Effect of Bazedoxifene and Conjugated Estrogen (Duavee) on Breast Cancer Risk Biomarkers in High-Risk Women: A Pilot Study. Cancer Prev Res (Phila). 2019 Oct;12(10):711-720. doi: 10.1158/1940-6207.CAPR-19-0315. Epub 2019 Aug 16. PMID 31420361